CLINICAL TRIAL: NCT07373522
Title: Biliary Stent For Management Of Esophageal Stricture In Children: A Randomized Controlled Trial.
Brief Title: Biliary Stent For Management Of Esophageal Stricture In Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ahmed Farag
Record Dates: First submitted 2026-01-20; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Esophageal Stenosis in Children

STUDY DESIGN:
Intervention Model Description: This study included children who were admitted to investigators' center to repair esophageal stricture. Cases were collected in the period from December 2025 to January 2026. the sample size was 40 patients divided into two equal groups. Group (1) included 20 patients managed by surgical intervention , group (2) included 15 patients managed by endoscopic intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic Group (Active Comparator): endoscopic stenting of esophageal stricture by fully covered self expanding metallic stent.
  Interventions: Procedure: endoscopic stenting of esophageal stricture by fully covered self expanding metallic stent
- surgical group (No Intervention): resection and reconstruction of stenosed esophageal segemt

INTERVENTIONS:
Procedure: endoscopic stenting of esophageal stricture by fully covered self expanding metallic stent — endoscopic stenting of esophageal stricture by fully covered self expanding metallic stent
  Arms: Endoscopic Group

SUMMARY:
All patients will subjected to the followings:

patients were selected by randomization method, full history taking, Complete physical examination, laboratory investigations (complete blood picture, liver and kidney functions, coagulation profile, tumor marker tests, serum electrolytes), patients were assessed radio-logically by abdominal x- ray , abdominal ultrasound, pelvic and abdominal CT.

For patients in EG, we began with assessment of the site & lenght of stricture . In this study, we used fully covered self expanded metallic biliary stent.

For patients in SG, we usually did gastrotomy feeding tube, excision and re-anastomosis, or did esophageal replacement surgery

DETAILED DESCRIPTION:
Technical design:

A- Site of the study: The investigators included all patients who were presented to General Surgery Department with Esophgeal Stricuture In Children at Zagazig University hospital between (December 2024 to December 2025).

B- Sample size:

c- Sample selection: Included patients were randomized at a 1:1 ratio to "Endoscopic Group, EG" or "Surgical Group , SG" via the drawing of sealed envelopes containing computer-generated random numbers prepared by a third party before the start of the intervention.(simple random sample).

D- Subjects: Patients will be divided into 2 groups in accordance type of preoperative

Therapy :

Group 1: "Endoscopic Group, EG" included patients. Group 2: "Surgical Group , SG" included patients.

Inclusion criteria:

Patients with Esophgeal Stricuture In Children , recurrent fistula , failued conservative meaures .patient with good general condition (ASA I&II).

Exclusion criteria:

We excluded patients who bad general condition (ASAIII&IV&V), respond to conservative measures.

E- Data collection (tools): All patients will subjected to the followings:

patients were selected by randomization method, full history taking, Complete physical examination, laboratory investigations (complete blood picture, liver and kidney functions, coagulation profile, tumor marker tests, serum electrolytes), patients were assessed radio-logically by abdominal x- ray , abdominal ultrasound, pelvic and abdominal CT.

Study design (operational study):

A. Type of the study : A randomized Controlled Trial.

B. Steps of performance:

1. Complete history taking.
2. Clinical and laboratory results.
3. Radiological results.
4. Endoscopic management of Esophgeal Stricuture In Children.
5. Analysis of the results.
6. Preparing conclusion and recommendation.

C-Study techniques (procedure):

For patients in EG, we began with assessment of the site & lenght of stricture . In this study, we used fully covered self expanded metallic biliary stent.

For patients in SG, we usually did gastrotomy feeding tube, excision and re-anastomosis, or did esophageal replacement surgery.

D-Outcomes:

Primary and secondary outcomes were incidence of postoperative hospital stay and complications in each group during the 3-months follow-up period, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Esophageal Stricture In Children.
* recurrent fistula.
* failed conservative measures .
* patient with good general condition (ASA I&II).

Exclusion Criteria:

* bad general condition (ASAIII&IV&V).
* respond to conservative measures.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
incidence of recurrence of stenosis | within one week after the endoscopy
  incidence of recurrence of stenosis

SECONDARY OUTCOMES:
incidence of side effects of endoscopy | within one month after the endoscopy
  incidence of side effects of endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Said Negm, Principal Investigator — Zagazig University Faculty Medicine
Locations (1):
- Zagazig University, Zagazig, Sharquia, Egypt

IPD SHARING:
Plan to Share IPD: No